CLINICAL TRIAL: NCT07016334
Title: The Role of Metabolic, Immune, and Neurotrophic Markers in the Etiology of Eating Disorders Using Neonatal Bloodspots
Brief Title: We Analyse Metabolites in Dried Blood Spots From Newborns That Later in Life Developed an Eating Disorder.
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ida AK Nilsson, Principal Investigator, Karolinska Institutet
Other Study IDs: Analysis of blood spots in ED
Record Dates: First submitted 2025-05-21; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 44 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anorexia nervosa: Diagnosed (life-time) with anorexia nervosa
- Bulimia nervosa: Diagnosed (life-time) with bulimia nervosa
- Controls: Never diagnosed with anorexia or bulimia nervosa

SUMMARY:
Anorexia nervosa (AN) and bulimia nervosa (BN) are serious eating disorders (EDs) with significant morbidity and mortality. Genetic studies have shown associations between EDs and metabolic traits, and longitudinal studies indicate distinct weight trajectories in children who later develop AN or BN, suggesting early involvement of metabolic factors. Biological studies also reveal differences in immune and neurotrophic markers in individuals with EDs compared to controls. Intriguingly, metabolites measured in neonatal blood could serve as very early markers of ED risk, unconfounded by state or scar factors related to prolonged starvation.

Here the investigators propose to comprehensively analyze neonatal biomarkers (metabolic, immune, and neurotrophic), epidemiological factors, and genetics to understand ED risk and develop risk prediction models

ELIGIBILITY:
Inclusion Criteria:

- in PKU-register with or withou life-time diagnosis of anorexia or bulimi nervosa

Exclusion Criteria:

* not in PKU register

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population born from 1981 with/or with out diagnosis of anorexia or bulimia nervosa
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Metabolomic factors measured by mass-spectrometry | Sampled at birth (day 1)
  Metabolomic factors such as amino acids, sugars, lipids, and organic acids extracted from dried blood spots sampled at birth are measured by mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden